CLINICAL TRIAL: NCT06897124
Title: Patients Experiences of Rehabilitation After Reverse Shoulder Arthroplasty - a Qualitative Interview Study
Brief Title: Patients Experiences of Rehabilitation Before and After Reverse Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: VGFOUSA-1020701
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: Reverse shoulder arthroplasty, qualitative research, physiotherapy, experiences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women and men, who had undergone surgery with reverse shoulder arthroplasty.: The participants were recruited from three different hospitals in Western Sweden: a local hospital, a county hospital, and a university hospital. The inclusion criteria encompassed patients who had undergone elective surgery involving reverse shoulder arthroplasty in the Västra Götaland region who demonstrated proficiency in both spoken and written Swedish.

SUMMARY:
Reverse shoulder arthroplasty is a complex surgical procedure requiring thorough rehabilitation, and its frequency is increasing globally. While previous studies have quantitatively examined postoperative outcomes, such as pain levels and shoulder function, no research has yet explored patients' subjective experiences of the rehabilitation process before and after surgery. Purpose of the study was to explore patients' experiences of undergoing reverse shoulder arthroplasty and the associated rehabilitation process.

DETAILED DESCRIPTION:
Surgery with total shoulder arthroplasty is a procedure that has increased in number in the last twenty years, and it is the third most common prosthetic surgery in the world after hip and knee. There are two types of shoulder arthroplasty, anatomical and reverse. When the rotator cuff is severely impaired or completely dysfunctional, a reverse shoulder prosthesis is used, in which the anatomical positions of the ball and socket are reversed.

There are thus several factors that the treating physiotherapist needs to take into account. Research on reverse shoulder arthroplasty has primarily focused on evaluations using quantitative measures. Qualitative research from the patient's perspective can provide a deeper understanding of their expectations and experiences, offering insights that complement and fill the gaps left by quantitative research. Gaining insight into patients' experiences would be valuable for physiotherapists working with this group, as it may help identify areas for improvement in care to better meet patients' needs.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria encompassed patients who had undergone elective surgery involving reverse shoulder arthroplasty in the Västra Götaland region who demonstrated proficiency in both spoken and written Swedish.

Exclusion Criteria:

Exclusion criteria applied to cases where the study leader had served as the patient's physiotherapist, the presence of neurological disorders, or the occurrence of surgical complications, such as infection or fracture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had undergone surgery with a reverse shoulder prosthesis during the period from September to November 2021. Based on background variables from the surgery lists, a strategic selection of participants was made to achieve variation in terms of gender, age, and geographic area.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
Patients' experiences of undergoing surgery and rehabilitation with reverse shoulder arthroplasty. | From time of surgery to end of rehabilitation, approximately 0-7,8 months.
  Qualitative semi structured individual in-depth interviews were analysed using qualitative content analysis. Fifteen persons, women and men, who had undergone surgery with reverse shoulder arthroplasty between six to twelve months previously, were recruited to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Larsson, RPT, PhD, Study Chair — Research, Education, Development & Innovation, Primary Health Care, Region Västra Götaland, Sweden.
Locations (1):
- Research, Education, Development & Innovation, Primary Health Care, Region Västra Götaland, Sweden, Alingsås, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No